CLINICAL TRIAL: NCT01221467
Title: An Open-label, Single-centre, Randomised, 2-period Cross-over Study to Assess the Efficacy, Safety and Utility of Real-time Continuous Subcutaneous Glucose Monitoring Combined With Overnight Closed-loop Glucose Control in the Home Setting in Comparison With Real-time Continuous Subcutaneous Glucose Monitoring Alone in Adolescents With Type 1 Diabetes on Subcutaneous Insulin Infusion Pump Therapy.
Brief Title: Closing the Loop in Youth With Type 1 Diabetes in the Home Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Principal Research Associate, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APCam06
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Overnight closed-loop combined with real-time CGM (Active Comparator)
  Interventions: Device: Overnight closed-loop
- Real-time CGM alone (Active Comparator)
  Interventions: Device: Overnight closed-loop

INTERVENTIONS:
Device: Overnight closed-loop — The closed-loop system is purpose-built and comprises a hand-held computer containing the algorithm and communicating with the CGM device and the insulin pump.

SUMMARY:
Type 1 diabetes (T1D) is one of the most common chronic childhood diseases requiring life-long insulin therapy. Children and adolescents with T1D need regular insulin injections or the continuous insulin delivery using an insulin pump in order to keep blood glucose levels normal. The investigators know that keeping blood sugars in the normal range will help prevent long-term diabetes-related complications involving the eyes, kidneys and heart. However, achieving treatment goals can be very difficult as the tighter the investigators try to control blood glucose levels, the greater the risk to develop symptoms and signs of low glucose levels (hypoglycaemia). This is a particular problem at night and one solution is to develop a system whereby the amount of insulin injected is controlled by a computer and is very closely matched to the blood sugar levels on a continuous basis. This can be achieved by what is known as a "closed-loop system" where a small glucose sensor placed under the skin communicates with a computer containing an algorithm that drives an insulin pump. The investigators have been testing such a system in Cambridge over the last three years in children and have found that this system is effective at preventing nocturnal hypoglycaemia. The next stage of this research is to test the system for a longer period of time at home. In the present study the investigators are planning to study 16 adolescents aged 12-18 years on insulin pump therapy. During 21 nights glucose will be controlled by the computer and during the other 21 nights the subjects will make their own adjustments to the insulin therapy. The investigators will then analyze the data to determine the effect of the computer algorithm in keeping glucose levels between 3.9 and 8 mmol/L (normal levels) and reducing the time they spent with glucose below 3.9 mmol/L (hypoglycaemia). Subjects' response to the use of the system in terms of life-style change, daily diabetes management and fear of hypoglycaemia will be assessed. The investigators will also test for longer term glucose control by measuring glycated haemoglobin and other blood parameters.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is between 12 and 18 years of age (inclusive)
2. The subject has type 1 diabetes, as defined by WHO for at least 1 year or is confirmed C-peptide negative
3. The subject will all have been insulin pump user for at least 3 months, with good knowledge of insulin self-adjustment as judged by the investigator
4. The subject willing to perform regular finger-prick blood glucose monitoring, with at least 4 blood glucose measurements taken every day
5. HbA1c ≤ 10 % based on analysis from central laboratory or equivalent
6. The subject is literate in English
7. Able to accommodate on site or in close proximity member(s) of study team for supervised closed-loop night(s)

Exclusion Criteria:

1. Non-type 1 diabetes mellitus including those secondary to chronic disease
2. Any other physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
3. Current treatment with drugs known to interfere with glucose metabolism, eg systemic corticosteroids, non-selective beta-blockers and MAO inhibitors etc
4. Known or suspected allergy against insulin
5. Subjects with clinical significant nephropathy, neuropathy or proliferative retinopathy as judged by the investigator
6. Total daily insulin dose ≥ 2 IU/kg/day
7. Pregnancy, planned pregnancy, or breast feeding
8. Prolonged use of any continuous glucose monitoring devices over the last 1 month prior the study
9. Severe visual impairment
10. Severe hearing impairment
11. Subjects using implanted internal pace-maker -

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Outcome | At least 7 days of valid CGM nights (midnight-7:30)
  The primary objective of the study is to assess the efficacy of continuous glucose monitoring (CGM) combined with overnight automated closed-loop glucose control in maintaining CGM glucose levels within the target range from 3.9 to 8.0 mmol/L, when compared with the use of CGM alone in the home setting.

SECONDARY OUTCOMES:
Secondary outcomes | At least 7 days of valid CGM nights (midnight-7:30)
  As a secondary research question, the safety of overnight automated closed-loop glucose control in terms of number of episodes of severe hypoglycaemia as well as the number of subjects experiencing severe hypoglycaemia and other adverse events.
  Furthermore, the frequency and duration of use of the closed-loop system will be evaluated. Subjects' perception in terms of life-style change, daily diabetes management and fear of hypoglycaemia will be assessed using questionnaires and a qualitative interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics, Weston paediatric diabetes centre, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Thabit H, Elleri D, Leelarathna L, Allen J, Lubina-Solomon A, Stadler M, Walkinshaw E, Iqbal A, Choudhary P, Wilinska M, Barnard K, Heller S, Amiel S, Evans M, Dunger D, Hovorka R. Unsupervised overnight closed loop insulin delivery during free living: analysis of randomised cross-over home studies in adults and adolescents with type 1 diabetes. Lancet. 2015 Feb 26;385 Suppl 1:S96. doi: 10.1016/S0140-6736(15)60411-1. PMID 26312919
- [Derived] Thabit H, Leelarathna L, Wilinska ME, Elleri D, Allen JM, Lubina-Solomon A, Walkinshaw E, Stadler M, Choudhary P, Mader JK, Dellweg S, Benesch C, Pieber TR, Arnolds S, Heller SR, Amiel SA, Dunger D, Evans ML, Hovorka R. Accuracy of Continuous Glucose Monitoring During Three Closed-Loop Home Studies Under Free-Living Conditions. Diabetes Technol Ther. 2015 Nov;17(11):801-7. doi: 10.1089/dia.2015.0062. Epub 2015 Aug 4. PMID 26241693
- [Derived] Hovorka R, Elleri D, Thabit H, Allen JM, Leelarathna L, El-Khairi R, Kumareswaran K, Caldwell K, Calhoun P, Kollman C, Murphy HR, Acerini CL, Wilinska ME, Nodale M, Dunger DB. Overnight closed-loop insulin delivery in young people with type 1 diabetes: a free-living, randomized clinical trial. Diabetes Care. 2014;37(5):1204-11. doi: 10.2337/dc13-2644. PMID 24757227